CLINICAL TRIAL: NCT07122063
Title: A Multicenter, Open-Label Phase I/II Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SYS6045 in Patients With HER2-Positive, Expressing, or Mutated Advanced Malignant Solid Tumors
Brief Title: Clinical Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SYS6045 in Patients With HER2-Positive, Expressing, or Mutated Advanced Malignant Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYS6045-001
Record Dates: First submitted 2025-07-23; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Eligible participants will receive SYS6045 via intravenous infusion on Day 1 of each treatment cycle. Cycles repeat every 3 weeks (Q3W, every 3 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYS6045 (Experimental): SYS6045,Q3W
  Interventions: Drug: SYS6045

INTERVENTIONS:
Drug: SYS6045 — SYS6045, IV Q3W

SUMMARY:
This study is the first-in-human (Phase I/II) trial of SYS6045, a multicenter, open-label, dose-escalation and dose-expansion clinical study. It aims to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary anti-tumor activity of SYS6045 in patients with HER2-positive, expressing, or mutated advanced solid tumors.

DETAILED DESCRIPTION:
The trial consists of two parts:Phase I (dose-escalation study): divided into two segments:Dose-escalation phase and PK expansion phase Phase II (dose-expansion study)

ELIGIBILITY:
Inclusion Criteria:

1. Age : ≥18 years.
2. ECOG Performance Status : 0-1.
3. Tumor Lesion Requirements:

   Dose Escalation Phase: At least one evaluable lesions per RECIST v1.1. PK Expansion Phase and Phase II (Dose Expansion Study): At least one measurable lesion per RECIST v1.1.
4. Life Expectancy: ≥3 months.
5. Adequate Organ Function (confirmed by laboratory tests within 14 days prior to enrollment, without transfusion or hematopoietic growth factor support):

   Absolute Neutrophil Count (ANC) ≥1.5×10⁹/L Platelet Count (PLT) ≥100×10⁹/L Hemoglobin (Hb) ≥90 g/L Total Bilirubin (TBIL) ≤1.5×ULN (≤3×ULN for participants with liver metastases or hepatocellular carcinoma) ALT/AST ≤2.5×ULN (≤5×ULN for participants with liver metastases or hepatocellular carcinoma) Serum Creatinine (Cr) <1.5×ULN Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN; International Normalized Ratio (INR) ≤1.5×ULN
6. Left Ventricular Ejection Fraction (LVEF): ≥50% during screening.
7. Fertile males or females must agree to use reliable contraceptive methods (hormonal contraceptives, barrier methods, or abstinence) with their partners during the trial and for ≥7 months after the last dose. Women of childbearing potential must have a negative blood pregnancy test within 7 days before enrollment.
8. Capable of understanding and voluntarily signing the informed consent form Additional Inclusion Criteria for Phase I (Dose Escalation Phase)
9. Histologically or cytologically confirmed advanced/unresectable, or metastatic solid tumors.
10. HER2-positive, HER2-expressing, or HER2-mutated advanced solid tumors confirmed by a local laboratory (excluding lung cancer; HER2 positivity in lung cancer requires central laboratory confirmation). Prior failure of ≥1 line of standard therapy required.

    Note: Standard therapy is defined as treatment according to established guidelines, consensus, or clinical practice standards. Treatment failure is defined as disease progression or tumor recurrence/metastasis during or after therapy.

    Additional Inclusion Criteria for Phase I (PK Expansion Phase)
11. Histologically or cytologically confirmed advanced/unresectable, or metastatic solid tumors.
12. HER2-aberrant, HER2-expressing, or HER2-mutated advanced solid tumors confirmed by a local laboratory (Note: For lung cancer, HER2 genetic alterations may be accepted based on local reports, subject to sponsor review and approval. HER2 IHC/FISH testing for lung cancer requires central laboratory confirmation).

    * Specific Criteria for Breast Cancer Cohort: Histologically or cytologically confirmed advanced/unresectable or metastatic breast cancer.
    * Advanced/unresectable or metastatic colorectal cancer: Histologically or cytologically confirmed, HER2-aberrant (including amplification, overexpression, or mutation).
    * Advanced/unresectable or metastatic non-small cell lung cancer (NSCLC): Histologically or cytologically confirmed, HER2-aberrant).

    Additional Inclusion Criteria for Phase II (Dose Expansion Study).
13. Documented disease progression or intolerance to the most recent systemic anti-tumor therapy based on radiological and/or pathological evidence.
14. HER2-positive, HER2-expressing, or HER2-mutated advanced solid tumors confirmed by a local laboratory (Note: For lung cancer, HER2 positivity requires central laboratory confirmation), with prior failure of at least one line of standard therapy.

    * Cohort 2a (HER2-positive breast cancer): Histologically or cytologically confirmed advanced/unresectable or metastatic breast cancer, with prior failure of ≥2 lines of standard therapy.
    * Cohort 2b (HER2-positive breast cancer): Histologically or cytologically confirmed advanced/unresectable or metastatic breast cancer, with prior failure of ≥1 line of standard therapy.
    * Cohort 2c (HER2-positive colorectal cancer): Histologically or cytologically confirmed advanced/unresectable or metastatic colorectal cancer.
    * Cohort 2d (HER2-positive non-small cell lung cancer, NSCLC): Histologically or cytologically confirmed advanced/unresectable or metastatic NSCLC.
    * Cohort 2e (Other solid tumors excluding above types): Histologically or cytologically confirmed advanced/unresectable or metastatic solid tumors (excluding breast, colorectal, and NSCLC), with HER2 expressionor HER2 mutation.

Exclusion Criteria:

1. Prior treatment with HER2-targeted ADC carrying a topoisomerase I inhibitor payload (e.g., DS-8201) or other TOP1 ADCs (Patients who received such agents in the neoadjuvant/adjuvant setting and experienced recurrence ≥12 months after treatment completion may be enrolled)[Applicable to: Phase I PK expansion and Phase II dose expansion studies].
2. Active neurological conditions, including: Spinal cord compression, clinically active brain metastases (untreated, symptomatic, or requiring corticosteroids/anticonvulsants for symptom control), carcinomatous meningitis or leptomeningeal disease. Asymptomatic CNS metastases with stable status ≥4 weeks after therapy and on tapering corticosteroids (≤10 mg/day prednisone equivalent) are allowed.
3. Chronic immunosuppressive therapy, including: Long-term immunosuppressants (e.g., cyclosporine),Systemic corticosteroids (>20 mg/day prednisone equivalent), Topical/nasal/inhaled corticosteroids are permitted.
4. Unresolved toxicities from prior anticancer therapy Not recovered to CTCAE v5.0 Grade ≤1 or baseline levels(Alopecia, hyperpigmentation, or isolated lab abnormalities deemed non-risky by the investigator).
5. Recent anticancer treatments (relative to first dose): Immunotherapy/macromolecular agents ≤4 weeks, Cytotoxic chemotherapy/small-molecule therapy ≤2 weeks, Traditional Chinese medicine ≤2 weeks.
6. Strong CYP3A4 inducers/inhibitors or OATP1B1/1B3 inhibitors≤2 weeks before first dose, or Within 5 half-lives (whichever is longer).
7. Major surgery or invasive procedures≤28 days before first dose Planned tumor resection during the study period.
8. Known severe allergies to any component of the investigational drug, History of severe hypersensitivity to monoclonal antibodies (e.g., trastuzumab) .
9. Active bacterial, fungal, or viral infections within 14 days prior to the first dose (Defined as requiring intravenous antimicrobial, antifungal, or antiviral therapy). Subjects without clinical manifestations of active infection prior to the first dose who are receiving prophylactic anti-infective treatment may be considered for enrollment.
10. Uncontrolled serous cavity effusions requiring frequent drainage or medical intervention within 7 days prior to the first dose, includes pleural, peritoneal, or pericardial effusions necessitating additional intervention within 2 weeks post-drainage (excluding acellular cytological testing of exudates)
11. History of immunodeficiency, including positive HIV antibody test.
12. Active HBV or HCV infection: Active HBV: HBsAg-positive with HBV DNA>2000 IU/mL，Active HCV: HCV-Ab-positive with HCV RNA>upper limit of normal (ULN).
13. History of non-infectious lung disease /pneumonitis requiring steroid therapy, current interstitial lung disease (ILD)/pneumonitis, or radiographically suspected ILD/pneumonitis during screening.
14. Severe cardiovascular disease history, including but not limited to:

    * Acute coronary syndrome within 6 months prior to the first dose.
    * Stroke or transient ischemic attack within 6 months prior to the first dose.
    * Pulmonary embolism or deep vein thrombosis within 3 months prior to the first dose.
    * Symptomatic heart failure of NYHA class ≥II.
    * Documented history of pulmonary embolism.
    * Prior myocardial infarction.
    * Pericarditis or pericardial effusion requiring clinical intervention.
    * Severe cardiac rhythm/conduction abnormalities (e.g., ventricular arrhythmias requiring intervention, grade II-III atrioventricular block).
    * QTcF>450 ms (male) or>470 ms (female), or history/family history of long QT syndrome.
    * Left ventricular ejection fraction (LVEF) <50%.
    * Uncontrolled hypertension (persistent SBP≥160 mmHg and/or DBP≥100 mmHg despite antihypertensive therapy) or poor adherence to antihypertensive medications
15. Pregnancy or lactation in female participants.
16. Presence of other conditions that may interfere with the subject's participation in study procedures, are not in the subject's best interest to participate, or may affect study outcomes: such as history of psychiatric disorders, substance abuse, or any other clinically significant diseases or conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 3 weeks
Incidence and severity of AEs | Up to 3 weeks
Recommended Phase II Dose (RP2D) | Up to 6 months
Objective Response Rate (ORR) | Up to 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  Assessed by investigators based on RECIST v1.1 criteria.
Disease Control Rate (DCR) | Up to 24 months
Progression-Free Survival (PFS) | Up to 24 months
  Assessed by investigators based on RECIST v1.1 criteria
Incidence and severity of AEs | Up to 24 months
Pharmacokinetic profile（AUC） | Up to 24 months
Rate of anti-SYS6045 antibodies (ADA) | Up to 24 months
Pharmacokinetic profile（Cmax） | Up to 24 months
Pharmacokinetic profile（Tmax） | Up to 24 months
Pharmacokinetic profile（t1/2） | Up to 24 months
Pharmacokinetic profile（CL） | Up to 24 months
Pharmacokinetic profile（MRT） | Up to 24 months
Rate of Neutralizing Antibodies (NAb)（if applicable） | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Juan Qu, doctor, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoing, China

IPD SHARING:
Plan to Share IPD: No